CLINICAL TRIAL: NCT03031353
Title: Misoprostol Before Elective Caesarean Section for Decreasing the Neonatal Respiratory Morbidity: A Randomized Controlled Trial
Brief Title: Misoprostol Before Elective Caesarean Section for Decreasing the Neonatal Respiratory Morbidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, Dr., Lecturer in obstertics and gynecology, Ain Shams University Hospital, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AinShamsU103
Record Dates: First submitted 2016-11-27; First posted 2017-01-25 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Transient Tachypnea Newborn; Cesarean Delivery Affecting Fetus
MeSH Terms: conditions — Transient Tachypnea of the Newborn | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): After preparing for elective caesarean section, the pessary will be given containing the misoprostol medication 1 hour before , women in the operating room, and the anaesthetic and surgical techniques will be standardized
  Interventions: Drug: Misoprostol
- Placebo (Active Comparator): After preparing for elective caesarean section, the pessary will be given containing placebo 1 hour before , women in the operating room, and the anaesthetic and surgical techniques will be standardized
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Misoprostol — Misoprostol is given before elective cesarean section as prophylaxis against post partum hemorrhage
  Other Names: Mesotac
  Arms: Misoprostol
Drug: Placebos — placebos tablet will be given before elective Cesarean sections
  Arms: Placebo

SUMMARY:
Neonatal respiratory distress may occur in either term or preterm newborns with a higher relative risk in preterm, and whether born vaginally or through caesarean section, but in a higher percentage after elective caesarean section whose rate is rising.

Prostaglandins may be given about one hour before an elective caesarean section after excluding the presence of contraindication to their use to decrease the neonatal respiratory diseases and thus, the number of children who suffered from bronchopulmonary dysplasia that occurs frequently in children who had previously TTN will diminish.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or more.
* Term singleton pregnancy (38 - 38+6 weeks gestation).
* Planned for elective transverse lower segment caesarean section with an indication.

Exclusion Criteria:

* Women with history of significant cardiac disease, eclampsia, pre eclampsia, epilepsy, severe asthma, severe allergic condition, vascular disease, renal or hepatic disease.
* Women with contraindication to prostaglandins as Glucoma or known hypersensitivity to prostaglandins or specifically for misoprostol.
* Psychological problem or mental disease that renders the patient not able to understand the nature, scope, and sequences of the study.
* Pregnancies with known foetal malformation/s or chromosomal aberration.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The need for admission to neonatal intensive care unit (NICU) | first 24 hours after delivery
  Number of newborns admitted to NICU for respiratory morbidity

SECONDARY OUTCOMES:
APGAR score below 6 at 5 minute | 5 minutes after delivery
  number of newborns delivered with APGAR score below 6 at 5 minutes

OTHER OUTCOMES:
neonatal mortality | first month after delivery
  number of neonates died from respiratory morbidity with one month of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No